CLINICAL TRIAL: NCT02476916
Title: A Phase 2, Open Label, Randomized, Dose Ranging, Safety, Efficacy, Pharmacokinetic and Pharmacodynamic Study of AG-348 in Adult Patients With Pyruvate Kinase Deficiency
Brief Title: A Study of AG-348 in Adult Participants With Pyruvate Kinase (PK) Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-003; 2015-000484-13 (EudraCT Number)
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pyruvate Kinase Deficiency
Keywords: Pyruvate Kinase Deficiency; Hemolytic anemia; Pyruvate Kinase Isoform R (PKR); Drive PK
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic | interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AG-348 50 mg BID (Experimental): Participants with PK deficiency received AG-348, 50 milligrams (mg), as initial dose, twice daily (BID) for the Core Period (Week 24).
  Interventions: Drug: AG-348
- AG-348 300 mg BID (Experimental): Participants with PK deficiency received AG-348, 300 mg, as initial dose, BID for the Core Period (Week 24).
  Interventions: Drug: AG-348

INTERVENTIONS:
Drug: AG-348 — Participants with PK deficiency were randomized to either receive AG-348, 50 or 300 mg, as initial doses, BID for the Core Period (Week 24). At the Week 24 visit, Core Period participants who had safely tolerated AG-348 and demonstrated clinical activity in response to AG-348 were potentially eligible to immediately roll over to the Extension Period for continued treatment. Participants were assigned to initial doses, however, over the course of the core period were treated across a range of doses due to treatment emergent adverse events (AEs) and hemoglobin (Hb) levels exceeding mid-point of sex-adjusted ranges.
  Other Names: Mitapivat

SUMMARY:
Study AG348-C-003 is a multicenter study designed to evaluate the safety and efficacy of different dose levels of AG-348 (mitapivat) in participants with PK deficiency.

DETAILED DESCRIPTION:
This is a Phase 2, open label, two arm, multicenter, randomized, dose-ranging study during which adult participants with PK deficiency will receive multiple doses of AG-348 for up to 24 weeks (Core Period); eligible participants may enter an Extension Period to receive AG-348 for up to 8 additional years. Data will be reviewed on a regular basis and study design, dose and schedule will be adapted based on these reviews. The study will evaluate the safety and tolerability of multiple doses of AG-348, pharmacokinetic and pharmacodynamic (PD) profile of AG-348 and early indicators of clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Male or female, aged 18 years and older
3. Known medical history of PK deficiency
4. PK deficiency confirmed by enzymatic assay at Screening
5. Genotypic characterization of PKR gene at Screening
6. Genotypic characterization of uridine-5'-diphosphate-glucuronyltransferase-A1 (UGTA1) gene to document underlying Gilbert's disease (Gilbert's disease patients are eligible)
7. Males Hb ≤ 12.0 g/dL, females Hb ≤ 11 g/dL
8. Transfusion independent, defined as no more than 3 units of red blood cells (RBC) transfused in 12 months prior to the first day of study dosing and no transfusions within 4 months of first day of study dosing
9. Splenectomized patients must have had the procedure at least 6 months prior to Screening and must be up-to-date in recommended vaccinations
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
11. Must be taking at least 1 mg folic acid daily in the 21 days prior to screening
12. Adequate organ function defined by liver function, kidney function, platelet count and coagulation assessments
13. Agreement to use approved contraceptive measures
14. Women must not be breastfeeding

    For entry into the Extension Period, patients must meet criteria # 15-16:
15. Must have completed 24 weeks of treatment during the Core Period and tolerated AG-348
16. The treating Investigator agrees that there is a potential for clinical benefit to continued treatment and recommends participation in the Extension Period and the Medical Monitor approves

Exclusion criteria

1. Hb ˃ 12.0 g/dL if male, Hb ˃11.0 g/dL if female
2. Additional diagnosis of other congenital or acquired blood disorder
3. Iron overload sufficiently severe to result in cardiac, hepatic or pancreatic insufficiency
4. Bone marrow or stem cell transplant
5. Clinically symptomatic cholelithiasis or cholecystitis
6. Currently enrolled in any other investigational trial. Participation in the PK Deficiency Natural History Study (NCT02053480) is permitted
7. Exposure to any investigational drug, device or procedure within 28 days prior to screening or during trial participation
8. Concurrent medical condition such as poorly controlled hypertension, heart failure, active infection, frequent post-splenectomy sepsis, Hepatitis B or C, Human Immunodeficiency Virus type 1 (HIV1) or Human Immunodeficiency Virus type 2 (HIV2) infection, poorly controlled diabetes mellitus, history of primary malignancy with the exception of curatively treated nonmelanomatous skin cancer, cervical cancer of breast cancer in situ
9. Major surgery in the last 6 months
10. Psychiatric disorder that could compromise the ability of the patient to cooperate with the study
11. Serum bilirubin higher to the upper limit of normal attributable to factors other than hemolysis or Gilbert's Syndrome
12. Use of restricted products known to strongly inhibit cytochrome P450 (CYP) 3A4 metabolism within 5 days prior to Prior Day 1 dosing, or to strongly induce cytochrome P450 3A4 (CYP3A4) metabolism within 28 days prior to Day 1 dosing, or to strongly inhibit P-glycoprotein transporter within 5 days prior to Day 1 dosing, or digoxin within 5 days prior to Day 1 dosing.
13. Heart-rate corrected QT interval - Fridericia's method (QTcF) interval ˃ 450 ms in male, QTcF > 470 ms in female, with the exception of patients with a left Bundle Branch Block
14. Cardiac arrhythmias that are clinically significant or treated with drugs that are substrates of CYP3A4
15. Allergy to sulfonamides if characterized by acute hemolytic anemia, anaphylaxis, rash of erythema multiforme type or Stevens-Johnson Syndrome
16. Any other medical or psychological condition deemed by the Investigator to be likely to interfere with a patient's ability to participate in the study
17. Patients will not be permitted to enter the Extension Period if: The patient experienced AEs during the Core Period that are considered by the treating Investigator or the Sponsor's designated Medical Monitor to pose a significant safety risk to the patient if treatment were to be extended

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2025-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - Stanford University, Palo Alto, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Wayne State University School of Medicine - Children's Hospital of Michigan, Detroit, Michigan
  - New York Presbyterian Hospital- Weil Cornell Medical College, New York, New York
  - Central Pennsylvania Clinic, Belleville, Pennsylvania
  - Children Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- University Health Network, Toronto, Ontario, Canada
- France (2):
  - Hôpital Saint-Vincent de Paul, Lille, Nord
  - Hôpital Henri Mondor, Créteil, Île-de-France Region
- UOC Oncoematologia Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grace RF, Rose C, Layton DM, Galacteros F, Barcellini W, Morton DH, van Beers EJ, Yaish H, Ravindranath Y, Kuo KHM, Sheth S, Kwiatkowski JL, Barbier AJ, Bodie S, Silver B, Hua L, Kung C, Hawkins P, Jouvin MH, Bowden C, Glader B. Safety and Efficacy of Mitapivat in Pyruvate Kinase Deficiency. N Engl J Med. 2019 Sep 5;381(10):933-944. doi: 10.1056/NEJMoa1902678. PMID 31483964
- [Derived] Al-Samkari H, Grace RF, Glenthoj A, Andres O, Barcellini W, Galacteros F, Kuo KHM, Layton DM, Morado Arias M, Viprakasit V, Dong Y, Tai F, Hawkins P, Gheuens S, Morales-Arias J, Gilroy KS, Porter JB, van Beers EJ. Early-onset reduced bone mineral density in patients with pyruvate kinase deficiency. Am J Hematol. 2023 Mar;98(3):E57-E60. doi: 10.1002/ajh.26830. Epub 2023 Jan 9. No abstract available. PMID 36594181
- [Derived] Rab MAE, Van Oirschot BA, Kosinski PA, Hixon J, Johnson K, Chubukov V, Dang L, Pasterkamp G, Van Straaten S, Van Solinge WW, Van Beers EJ, Kung C, Van Wijk R. AG-348 (Mitapivat), an allosteric activator of red blood cell pyruvate kinase, increases enzymatic activity, protein stability, and ATP levels over a broad range of PKLR genotypes. Haematologica. 2021 Jan 1;106(1):238-249. doi: 10.3324/haematol.2019.238865. PMID 31974203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the core period of the study at 14 investigative sites in the 6 countries from 13 July 2015 to 14 July 2017 (data cut-off date). The core period is completed, and results of this period are reported. The extension period is ongoing.
Pre-assignment Details: A total of 52 participants were enrolled in the Core Period of the study. Out of 52 participants, 9 discontinued during the core period, and 43 completed the core period. Out of these 43, 36 entered the extension period, and 7 did not enter the extension period and were followed up to 4 weeks after their last dose of AG-348 in the core study.
Groups:
- AG-348 50 mg BID: Participants with Pyruvate Kinase (PK) deficiency received AG-348, 50 milligrams (mg), as initial dose, twice daily (BID) for 24 weeks (Core Period). Participants were assigned to initial doses, however, over the course of the Core Period were treated across a range of doses due to treatment emergent adverse events (AEs) and hemoglobin (Hb) levels exceeding mid-point of sex-adjusted ranges. At the Week 24 visit, Core Period participants who had safely tolerated AG-348 and demonstrated clinical activity in response to AG-348 were potentially eligible to immediately roll over to the Extension Period for continued treatment. If participants chose not to enroll, they were followed up to four weeks after the last dose of AG-348.
- AG-348 300 mg BID: Participants with PK deficiency received AG-348, 300 mg, as initial dose, BID for 24 weeks (Core Period). Participants were assigned to initial doses, however, over the course of the Core Period were treated across a range of doses due to treatment emergent AEs and Hb levels exceeding mid-point of sex-adjusted ranges. At the Week 24 visit, Core Period participants who had safely tolerated AG-348 and demonstrated clinical activity in response to AG-348 were potentially eligible to immediately roll over to the Extension Period for continued treatment. If participants chose not to enroll, they were followed up to four weeks after the last dose of AG-348.
Period: Core Period
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Started | 27 | 25
Completed | 21 | 22
Not Completed | 6 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Investigator decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Period: Extension Period
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Started (A total of 36 participants who had clinical activity and tolerated dose entered Extension Period.) | 18 | 18
Completed | 0 | 0
Not Completed | 18 | 18
Not completed — Prematurely Discontinued Treatment | 6 | 1
Not completed — On Treatment | 12 | 17

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who had received at least one dose of study drug.
Groups:
- AG-348 50 mg BID: Participants with PK deficiency received AG-348, 50 mg, as initial dose, BID for 24 weeks (Core Period). Participants were assigned to initial doses, however, over the course of the Core Period were treated across a range of doses due to treatment emergent AEs and Hb levels exceeding mid-point of sex-adjusted ranges. At the Week 24 visit, Core Period participants who had safely tolerated AG-348 and demonstrated clinical activity in response to AG-348 were potentially eligible to immediately roll over to the Extension Period for continued treatment. If participants chose not to enroll, they were followed up to four weeks after the last dose of AG-348.
- Total: Total of all reporting groups
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (11.26) | 37.7 (12.03) | 34.1 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 18 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 21 | 43
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AEs) in the Core Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered study drug-related.
Time Frame: Up to Week 24
Population: The Safety Analysis Set included all participants who had received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
percentage of participants | 96.3 | 100.0

2. Secondary Outcome: Percentage of Participants Experiencing at Least One AE Over the Duration of the Extension Period
Description: as for outcome 1
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Hemoglobin (Hb) Value at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Increased Hb values indicate improvement.
Time Frame: Baseline and Week 24
Population: The Efficacy Analysis Set included all participants who enrolled and received any study treatment for at least 3 weeks. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
grams per deciliter (g/dL)
  Baseline | 9.243 (1.4757) | 8.636 (1.1664)
  Change at Week 24: number analyzed (Participants) | 23 | 24
  Change at Week 24 | 1.205 (1.4181) | 1.611 (1.7058)

4. Secondary Outcome: Change From Baseline in Hb Value Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Increased Hb values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Hematocrit at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Increased hematocrit values indicate improvement.
Time Frame: Baseline and Week 24
Population: The Safety Analysis Set included all participants who had received at least one dose of study drug. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: volume per volume (V/V)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
volume per volume (V/V)
  Baseline | 0.289 (0.0470) | 0.268 (0.0367)
  Change at Week 24: number analyzed (Participants) | 23 | 23
  Change at Week 24 | 0.033 (0.0414) | 0.045 (0.0499)

6. Secondary Outcome: Change From Baseline in Hematocrit Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Increased hematocrit values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in Reticulocyte Count at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased reticulocyte count values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cells * 10^9/liter
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
cells * 10^9/liter
  Baseline | 493.248 (234.2242) | 549.436 (291.5301)
  Change at Week 24: number analyzed (Participants) | 23 | 23
  Change at Week 24 | -99.248 (309.9473) | -46.222 (351.9823)

8. Secondary Outcome: Change From Baseline in Reticulocyte Count Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased reticulocyte count values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in Haptoglobin at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Increased haptoglobin values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
gram per liter (g/L)
  Baseline: number analyzed (Participants) | 24 | 25
  Baseline | 0.246 (0.1474) | 0.240 (0.2082)
  Change at Week 24: number analyzed (Participants) | 18 | 23
  Change at Week 24 | 0.128 (0.2845) | 0.139 (0.2726)

10. Secondary Outcome: Change From Baseline in Haptoglobin Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Increased haptoglobin values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline in Carbon Monoxide at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased carbon monoxide values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage Hb bound to carbon monoxide
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
percentage Hb bound to carbon monoxide
  Baseline: number analyzed (Participants) | 19 | 20
  Baseline | 5.263 (1.7270) | 6.200 (2.3079)
  Change at Week 24: number analyzed (Participants) | 16 | 17
  Change at Week 24 | -1.063 (2.2940) | -1.706 (3.2742)

12. Secondary Outcome: Change From Baseline in Carbon Monoxide Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased carbon monoxide values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

13. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH) at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased LDH values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
units per liter (U/L)
  Baseline | 282.074 (188.3558) | 254.840 (122.3587)
  Change at Week 24: number analyzed (Participants) | 24 | 23
  Change at Week 24 | -26.292 (145.3151) | -8.913 (139.8509)

14. Secondary Outcome: Change From Baseline in LDH Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased LDH values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

15. Secondary Outcome: Change From Baseline in Total Bilirubin at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased total bilirubin values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
milligrams per deciliter (mg/dL)
  Baseline | 5.152 (2.3407) | 5.608 (3.4625)
  Change at Week 24: number analyzed (Participants) | 24 | 24
  Change at Week 24 | -1.921 (1.9465) | -3.017 (2.5848)

16. Secondary Outcome: Change From Baseline in Total Bilirubin Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased total bilirubin values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

17. Secondary Outcome: Change From Baseline in Indirect Bilirubin at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased indirect bilirubin values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
mg/dL
  Baseline | 4.752 (2.3629) | 5.208 (3.4272)
  Change at Week 24: number analyzed (Participants) | 24 | 22
  Change at Week 24 | -1.967 (1.8318) | -3.195 (2.5537)

18. Secondary Outcome: Change From Baseline in Indirect Bilirubin Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased indirect bilirubin values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

19. Secondary Outcome: Change From Baseline in Erythropoietin (EPO) at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased EPO values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
international units per liter (IU/L)
  Baseline | 85.448 (159.4090) | 60.900 (19.5188)
  Change at Week 24: number analyzed (Participants) | 24 | 24
  Change at Week 24 | -7.738 (33.1934) | -13.675 (26.5065)

20. Secondary Outcome: Change From Baseline in EPO Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased EPO values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

21. Secondary Outcome: Change From Baseline in Hepcidin at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased hepcidin values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
nanomoles per liter (nmol/L)
  Baseline: number analyzed (Participants) | 6 | 4
  Baseline | 3.392 (3.4013) | 4.988 (4.0416)
  Change at Week 24: number analyzed (Participants) | 4 | 3
  Change at Week 24 | 0.095 (1.4795) | -2.310 (2.5061)

22. Secondary Outcome: Change From Baseline in Hepcidin Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased hepcidin values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

23. Secondary Outcome: Change From Baseline in Ferritin at Week 24
Description: Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased ferritin values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
ng/mL
  Baseline | 860.852 (682.6346) | 859.680 (490.2734)
  Change at Week 24: number analyzed (Participants) | 24 | 23
  Change at Week 24 | 68.875 (388.1866) | -37.870 (308.0896)

24. Secondary Outcome: Change From Baseline in Ferritin Over the Duration of the Extension Period
Description: Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased ferritin values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

25. Secondary Outcome: Change From Baseline in Transferrin Saturation at Week 24
Description: Transferrin saturation is the ratio of serum iron to iron-binding capacity. Change (absolute change) from baseline was calculated as post-baseline value - baseline value. Decreased transferrin saturation values indicate improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 27 | 25
percentage of saturation
  Baseline: number analyzed (Participants) | 21 | 24
  Baseline | 50.143 (23.7388) | 64.292 (22.0779)
  Change at Week 24: number analyzed (Participants) | 16 | 20
  Change at Week 24 | -3.625 (16.1777) | -5.750 (19.8968)

26. Secondary Outcome: Change From Baseline in Transferrin Saturation Over the Duration of the Extension Period
Description: Transferrin saturation is the ratio of serum iron to iron-binding capacity. Change (absolute change) from baseline will be calculated as post-baseline value - baseline value. Decreased transferrin saturation values indicate improvement.
Time Frame: Up to approximately 8.5 years
Reporting Status: Not Posted

27. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Non-zero Concentration (AUC0-t) for AG-348 and Its Metabolite AGI-8702
Description: Pre-dose pharmacokinetic concentrations, if any, were excluded from the pharmacokinetic analyses.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose Day 1 and pre-dose, 0.5, 1, 2, 4, 8 hours post-dose Day 15
Population: The Pharmacokinetic Analysis Set included all participants from Core Period, without major protocol violation, who were enrolled and received any dose of study treatment, with sufficient plasma sample or whole blood data to assess pharmacokinetic parameters. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(hr*ng/mL)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 5 | 7
nanograms*hours per milliliter(hr*ng/mL)
  Day 1: AG-348 | 3287 (20.9) | 27930 (38.1)
  Day 15: AG-348: number analyzed (Participants) | 5 | 5
  Day 15: AG-348 | 3609 (38.2) | 11610 (11.3)
  Day 1: AGI-8702 | 235.6 (32.6) | 2637 (34.9)
  Day 15: AGI-8702: number analyzed (Participants) | 5 | 5
  Day 15: AGI-8702 | 425.8 (21.8) | 2235 (19.4)

28. Secondary Outcome: Maximum Plasma Concentration (Cmax) for AG-348 and Its Metabolite AGI-8702
Description: Pre-dose pharmacokinetic concentrations, if any, were excluded from the pharmacokinetic analyses.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose Day 1 and pre-dose, 0.5, 1, 2, 4, 8 hours post-dose Day 15
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- AG-348 300 mg: Participants with PK deficiency received AG-348, 300 mg, as initial dose, BID for 24 weeks (Core Period). Participants were assigned to initial doses, however, over the course of the Core Period were treated across a range of doses due to treatment emergent AEs and Hb levels exceeding mid-point of sex-adjusted ranges. At the Week 24 visit, Core Period participants who had safely tolerated AG-348 and demonstrated clinical activity in response to AG-348 were potentially eligible to immediately roll over to the Extension Period for continued treatment. If participants chose not to enroll, they were followed up to four weeks after the last dose of AG-348.
Arm/Group | AG-348 50 mg BID | AG-348 300 mg
Number analyzed (Participants) | 5 | 7
nanograms per milliliter (ng/mL)
  Day 1: AG-348 | 870.0 (9.2) | 7606 (41.8)
  Day 15: AG-348: number analyzed (Participants) | 5 | 5
  Day 15: AG-348 | 943.4 (30.7) | 5259 (35.6)
  Day 1: AGI-8702 | 41.03 (43.6) | 414.7 (35.6)
  Day 15: AGI-8702: number analyzed (Participants) | 5 | 5
  Day 15: AGI-8702 | 71.94 (22.0) | 533.7 (25.6)

29. Secondary Outcome: Time to Reach Peak Plasma Concentration (Tmax) for AG-348 and Its Metabolite AGI-8702
Description: Pre-dose pharmacokinetic concentrations, if any, were excluded from the pharmacokinetic analyses.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose Day 1 and pre-dose, 0.5, 1, 2, 4, 8 hours post-dose Day 15
Population: as for outcome 27
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 5 | 7
hour (hr)
  Day 1: AG-348 | 1.92 [0.97 to 2.03] | 1.97 [1.00 to 2.08]
  Day 15: AG-348: number analyzed (Participants) | 5 | 5
  Day 15: AG-348 | 1.00 [0.97 to 1.90] | 1.00 [0.42 to 2.00]
  Day 1: AGI-8702 | 2.00 [1.92 to 2.03] | 1.97 [1.00 to 2.13]
  Day 15: AGI-8702: number analyzed (Participants) | 5 | 5
  Day 15: AGI-8702 | 2.00 [1.95 to 4.00] | 1.00 [0.93 to 4.00]

30. Secondary Outcome: Apparent Clearance at Steady-State (Clss/F) for AG-348 and Its Metabolite AGI-8702
Description: Pre-dose pharmacokinetic concentrations, if any, were excluded from the pharmacokinetic analyses.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8 hours post-dose Day 15
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 5 | 7
liter per hour (L/hr)
  Day 15: AG-348: number analyzed (Participants) | 5 | 5
  Day 15: AG-348 | 12.27 (40.3) | 25.31 (11.7)
  Day 15: AGI-8702: number analyzed (Participants) | 3 | 3
  Day 15: AGI-8702 | 91.50 (31.0) | 128.2 (18.8)

31. Secondary Outcome: Maximum Change From Baseline Response Value Over 12 Hours Post-dose (BRmax) for Adenosine Triphosphate (ATP)
Description: Pre-dose concentration observed on Day 1 was used as Baseline for calculation of change from baseline.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose Day 1 and pre-dose, 0.5, 1, 2, 4, 8 hours post-dose Day 15
Population: The Pharmacodynamic (PD) Analysis Set included all participants from Core Period, without major protocol violation, who were enrolled and received any dose of study treatment, with sufficient plasma sample or whole blood data to assess PD parameters. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 5 | 7
µg/mL
  Change at Day 1: number analyzed (Participants) | 4 | 6
  Change at Day 1 | 16.50 (11.790) | 20.67 (6.8896)
  Change at Day 15: number analyzed (Participants) | 4 | 4
  Change at Day 15 | 1.500 (31.032) | 45.50 (60.995)

32. Secondary Outcome: Maximum Change From Baseline Response Value Over 12 Hours Post-dose (BRmax) for 2,3 - Diphosphoglycerate (2,3-DPG)
Description: Pre-dose concentration observed on Day 1 was used as Baseline for calculation of change from baseline.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose Day 1 and pre-dose, 0.5, 1, 2, 4, 8 hours post-dose Day 15
Population: The PD Analysis Set included all participants from Core Period, without major protocol violation, who were enrolled and received any dose of study treatment, with sufficient plasma sample or whole blood data to assess PD parameters. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/mL)
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
Number analyzed (Participants) | 5 | 7
microgram per milliliter (µg/mL)
  Change at Day 1: number analyzed (Participants) | 4 | 7
  Change at Day 1 | 42.25 (38.836) | 59.57 (58.569)
  Change at Day 15: number analyzed (Participants) | 4 | 5
  Change at Day 15 | -65.50 (69.745) | 8.200 (195.13)

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: The Safety Analysis Set included all participants who had received at least one dose of study drug.
Arm/Group | AG-348 50 mg BID | AG-348 300 mg BID
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 5/27 | 3/25
Other Adverse Events (participants affected / at risk) | 26/27 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-348 50 mg BID (N=27) | AG-348 300 mg BID (N=25)
Pharyngitis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AG-348 50 mg BID (N=27) | AG-348 300 mg BID (N=25)
Nausea (Gastrointestinal disorders) | 10 | 10
Vomiting (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Headache (Nervous system disorders) | 9 | 14
Dizziness (Nervous system disorders) | 5 | 2
Dysgeusia (Nervous system disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 7 | 2
Influenza (Infections and infestations) | 6 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Insomnia (Psychiatric disorders) | 5 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Fatigue (General disorders) | 4 | 4
Pyrexia (General disorders) | 1 | 5
Chest discomfort (General disorders) | 1 | 4
Asthenia (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 3
Hot flush (Vascular disorders) | 2 | 7
Flushing (Vascular disorders) | 2 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Palpitations (Cardiac disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained from the clinical study will be used towards the development of AG-348 and may be disclosed to regulatory authority(ies), other Investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT02476916/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02476916/SAP_001.pdf